CLINICAL TRIAL: NCT03584139
Title: IRIS Hook Assisted Phacoemulsification in Vitrectomized Eyes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Second Affiliated Hospital of Xi'an Jiaotong University (Other)
Responsible Party: Principal Investigator, Bai Ling, Associated Professor, Second Affiliated Hospital of Xi'an Jiaotong University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRIS hook
Record Dates: First submitted 2018-05-21; First posted 2018-07-12 (Actual); Last update posted 2020-03-06 (Actual); Status verified 2020-03

CONDITIONS: Cataract; Vitrectomy
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IRIS HOOK (Experimental): iris hook assisted maneuver in phacoemulsification
  Interventions: Device: IRIS HOOK
- TRADITION (Active Comparator): traditional phacoemulsification or phacoemulsification with 25-gauge vitreous irrigation
  Interventions: Device: TRADITION

INTERVENTIONS:
Device: IRIS HOOK — iris hook assisted maneuver in phacoemulsification
  Arms: IRIS HOOK
Device: TRADITION — traditional phacoemulsification or phacoemulsification with 25-gauge vitreous irrigation
  Arms: TRADITION

SUMMARY:
Although phacoemulsification in previously vitrectomized eyes is a relatively safe procedure comparing with extracapsular cataract surgery, it is still more challenging than in eyes without previous vitrectomy because of the anatomical differences after PPV. Intraoperative difficulties such as abnormal anterior chamber deepening, unstable posterior capsules, and weakened zonules have been reported.

The investigators aim to evaluate the efficacy and safety of a new simple iris hook assisted maneuver in phacoemulsification, then compare the incidence of intraoperative and postoperative complications of this technique with traditional phacoemulsification and phacoemulsification with 25-gauge vitreous irrigation. The latter two surgery methods are currently popular for cataract in vitrectomized eyes.

DETAILED DESCRIPTION:
With the continuous evolution in vitrectomy techniques and instrumentation, an increasing number of vitreorential disorders are being successfully managed with pars plana vitrectomy (PPV). Cataract is one of the most common complications seen in phakic patients following PPV, and the incidence of it ranges from 4 to 80%, even up to 100% in various studies.

Although phacoemulsification in previously vitrectomized eyes is a relatively safe procedure comparing with extracapsular cataract surgery, it is still more challenging than in eyes without previous vitrectomy because of the anatomical differences after PPV. Intraoperative difficulties such as abnormal anterior chamber deepening, unstable posterior capsules, and weakened zonules have been reported.

The investigators aim to evaluate the efficacy and safety of a new simple iris hook assisted maneuver in phacoemulsification, then compare the incidence of intraoperative and postoperative complications of this technique with traditional phacoemulsification and phacoemulsification with 25-gauge vitreous irrigation. The latter two surgery methods are currently popular for cataract in vitrectomized eyes.

ELIGIBILITY:
Inclusion Criteria:

1. patients with visually significant cataract following PPV
2. After PPV vitreous substitutes were air / gas (Perfluoropropane:C3F8) or BSS,
3. After PPV if vitreous substitute was silicone oil, that should be removed at least 3 months.
4. The duration between PPV / silicone oil remove and phacoemulsification should more than 3 months
5. Willing and able to comply with clinic visits and study-related procedures
6. Provide signed informed consent

Exclusion Criteria:

1. Eyes with a history of acute angle-closure glaucoma, trauma,
2. Eyes with a clinically dislocated or subluxated lens.
3. Active ocular or periocular infection in the study eye
4. Uncontrolled Blood Pressure
5. Pregnant or breast-feeding women
6. Participation in another simultaneous medical investigator or trial

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Stability of anterior chamber and pupil | Intraoperative
  The traditional phacoemulsification in vitrectomized eyes usually with more Intraoperative difficulties such as abnormal anterior chamber deepening and unstable pupil. To evaluate whether the new method will increase the stability of anterior chamber and pupil.
Time of operation | Intraoperative
  To evaluate whether the new method will shorten the operation time
Cumulative dissipated energy (CDE) | Intraoperative
  To evaluate whether the new method will decrease CDE. CDE reflect the damage of phacoemulsification to the eye, It can be acquired automatically from the phacoemulsification machine. The unit of CDE is mJ.

SECONDARY OUTCOMES:
The presence of intraoperative complications | Intraoperative
  The incidence of complications, including infusion deprivation syndrome, anterior capsulorhexis extension, iris trauma, descemets detachment, posterior capsular defect, nucleus drop, etc
Visual acuity (VA) | 3 months after opreation
  To evaluate whether the surgery can effectively increase VA.
Intraocular pressure(IOP) | 3 months after opreation
  The traditional phacoemulsification in vitrectomized eyes usually cause low IOP in the early stage, and sometimes induce detachment of choroid. To evaluate whether the new method will avoid the low IOP in the early stage.
The presence of postoperative complications | 3 months after opreation
  The incidence of complications, including corneal edema, cystoid macular edema, etc.

CONTACTS AND LOCATIONS:
Overall Officials: Ling Bai, MD,PhD, Principal Investigator — Second affiliated hospital of Xian Jiaotong University
Locations (1):
- Department of Ophthalmology, Second affiliated hospital of Xian Jiaotong University, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: No